CLINICAL TRIAL: NCT03821285
Title: Evaluation of Respiratory Function in Patients With Post-tuberculosis Lung Impairment After Pulmonary Tuberculosis Treatment or After Spontaneous Healing
Brief Title: Respiratory Function in Patients With Post-tuberculosis Lung Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università degli Studi dell'Insubria (Other)
Collaborators: Fondazione Salvatore Maugeri (Other); Azienda Ospedaliero Universitaria di Sassari (Other); Instituto Nacional de Enfermedades Respiratorias (Other Government)
Responsible Party: Principal Investigator, Dina Visca, Principal Investigator, Università degli Studi dell'Insubria
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2215CE
Record Dates: First submitted 2019-01-14; First posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Lung Diseases, Obstructive; Pulmonary Rehabilitation; Lung TB
Keywords: TB; Pulmonary rehabilitation; Lung function
MeSH Terms: conditions — Lung Diseases, Obstructive; Tuberculosis, Pulmonary

STUDY DESIGN:
Intervention Model Description: Prospective, multicentre international
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pulmonary rehabilitation (Experimental): Pulmonary rehabilitation program
  Interventions: Procedure: Pulmonary Rehabilitation

INTERVENTIONS:
Procedure: Pulmonary Rehabilitation — Pulmonary rehabilitation programme:15 aerobic-training sessions, 15 strength-training sessions for peripheral muscles, 3 face to face and/or Group educational sessions, if needed airways clearance techniques and/or inspiratory muscles training

SUMMARY:
Pulmonary tuberculosis (TB) is an important risk factor for chronic respiratory disease due to residual lung damage. A recent review of the literature on TB sequelae and rehabilitation has provided clear evidence that TB is definitively responsible for lung function impairment. Functional evaluation of TB patients after completion of pulmonary tuberculosis treatment or spontaneous healing should be considered as part of clinical care. Unfortunately, few studies are available in the literature investigating the physiopathology of lung damage, its impact on quality of life, the potential need for pulmonary rehabilitation (PR), and the effects of a PR program.Objectives of this prospective multicentre international study are: Primary Objective-to assess the exercise capacity 6-min walking test in patients with post-TB lung impairment after completion of pulmonary tuberculosis treatment or after spontaneous healing. Secondary Objectives-to assess the effects of the PR program on dyspnoea symptoms and muscle fatigue, quality of life.

DETAILED DESCRIPTION:
Methods Respiratory functional parameters at baseline and at the end of the 15 sessions rehabilitation programme (RP) will be collected at the participating Centre. Follow-up visit 1 year after completion of RP Baseline assessment

1. After signature of the informed consent to the study, patients will undergo a Pre-screening Visit: data on medical history, current pharmacological therapies, smoking (pack/year), vaccinations, physical examination, vital parameters (blood pressure, heart rate, respiratory rate, oxygen saturation in arterial blood), co-morbidities and Mini Mental State Examination will be collected.
2. Screening Visit (before the RP), during the visit the following data will be collected: number of TB disease episodes, detailed data on the last TB episode (age at onset of TB symptoms, age at TB diagnosis, anti-TB treatment duration, anti-TB drugs administered, socio-economic conditions, education level, physical examination, vital parameters, oxygen saturation in arterial blood, heart rate and respiratory rate). Pulmonary rehabilitation program tailored according to specific patient's needs.
3. Baseline assessment of respiratory function: arterial blood gas (ABG) analysis, spirometry, diffusing capacity of the lungs for carbon monoxide (DLCO), overnight oximetry, electrocardiogram (ECG), chest X-ray (CXR), High-resolution computed tomography (HRCT)
4. Assessment of the rehabilitation programme: functional evaluation (6MWT), muscle strength evaluation (five-repetition sit-to-stand test (5STS)), respiratory muscle strength (maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP)), symptoms evaluation (Dyspnea: Medical Research Council Questionnaire (MRC), Modified Borg pre/post 6MWT, Baseline and Transition Dyspnea Indexes (BDI-TDI) and Fatigue: Modified Borg pre/post 6MWT)
5. Assessment of the Quality of Life (QoL): CAT and St George's Respiratory Questionnaire.

Final assessment:

A final assessment will be done at the end of the rehabilitation programme and will include:

c) Only ABG, spirometry and DLCO d) and e).

Pulmonary rehabilitation programme

PR programme will include:

At least 15 aerobic-training sessions by cycle ergometer supervised by a respiratory therapist (5 session per week, 30 minutes each: 5 minutes warm up, 20 minutes training and 5 minutes warm-down) at constant load (calculated with Hill equation, Hill K, et al. Estimating maximum work rate during incremental cycle ergometry testing from six-minute walk distance in patients with chronic obstructive pulmonary disease. Arch Phys Med Rehabil. 2008;89(9):1782-7.) with an adherence of at least 80%.

1. At least 15 strength-training sessions for peripheral muscles (30 minutes calisthenics exercise) with an adherence of at least 80%.
2. At least 3 face to face and/or group educational sessions, for:

   * Optimization of inhalation techniques
   * Exercise training and maintenance programs
   * Daily physical activity
   * Airways clearance techniques
   * Long oxygen therapy home management.
3. According to individual needs, the PR program should include:

   * airways clearance techniques
   * inspiratory muscles training (with Threshold®)

Monitoring Anonymous data will be collected in a common electronic format (excel database).

Adverse events (AEs) and severe adverse events (SAEs) will be reported and registered.

Follow-up

Follow-up visit 1 year after completion of RP will include:

c) Only ABG, spirometry, DLCO and overnight oximetry d) and e) Statistical analysis A two-tailed p-value less than 0.05 will be considered statistically significant.

Qualitative and quantitative variables will be described with absolute and relative (percentages) frequencies and means (standard deviations -SD) or medians (interquartile ranges -IQR) depending on their normality, respectively. The mean difference between the two study groups in the 6MWT will be evaluated using the Student's t-test. Differences in the variables associated to the secondary objectives will be evaluated using the Chi-square or Student's t-test for qualitative and quantitative variables. A two-tailed p-value less than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

- Patients with post-TB lung impairment after completion of pulmonary tuberculosis treatment - Patients with post- TB impairment after spontaneous healing

Exclusion Criteria:

* Any unstable medical condition
* Musculoskeletal disorders contraindicating participation in the PR program
* Cognitive impairment (Mini Mental State Examination <22)
* Unable to sign informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-02-14 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2021-01-14 (Estimated)

PRIMARY OUTCOMES:
6-min walking test | 1 year
  Exercise capacity

SECONDARY OUTCOMES:
dyspnoea | 1 year
  Modified BORG scale (0-10) 0 better, 10 worse
muscle fatigue | 1 year
  Modified Borg scale (0-10) 0 better, 10 worse
health related quality of life | 1 year
  st. George Respiratory Questionnaire 0 better, 100 worse
health status | 1 year
  COPD Assessment test-CAT (0-40) 0 better, 40 worse

CONTACTS AND LOCATIONS:
Overall Officials: Giovan Battista Migliori, Prof, Study Director — ICS Maugeri, IRCCS
Locations (1):
- ICS Maugeri, IRCCS, Tradate, Varese, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tiberi S, Munoz-Torrico M, Duarte R, Dalcolmo M, D'Ambrosio L, Migliori GB. New drugs and perspectives for new anti-tuberculosis regimens. Pulmonology. 2018 Mar-Apr;24(2):86-98. doi: 10.1016/j.rppnen.2017.10.009. Epub 2018 Feb 24. PMID 29487031
- [Result] Munoz-Torrico M, Rendon A, Centis R, D'Ambrosio L, Fuentes Z, Torres-Duque C, Mello F, Dalcolmo M, Perez-Padilla R, Spanevello A, Migliori GB. Is there a rationale for pulmonary rehabilitation following successful chemotherapy for tuberculosis? J Bras Pneumol. 2016 Sep-Oct;42(5):374-385. doi: 10.1590/S1806-37562016000000226. PMID 27812638